CLINICAL TRIAL: NCT03457974
Title: Saliva Profiles in Children With Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Figen Seymen (Unknown); Merve Bayram (Unknown); Ezel Uslu (Unknown); Sule Batu (Unknown); Yegane Güven (Unknown)
Responsible Party: Principal Investigator, Mine Koruyucu, Principal Investigator, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2010/1109-378
Record Dates: First submitted 2018-02-23; First posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Cardiac Disease; Dental Caries
Keywords: saliva composition; antioxidant activity; caries risk factors; congenital cardiac disease
MeSH Terms: conditions — Heart Diseases; Dental Caries

STUDY DESIGN:
Intervention Model Description: cross sectional study was carried out with 42 CHD and 42 healthy children
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- congenital heart disease (Experimental): 42 patients
  Interventions: Other: saliva
- helathy children (Other): 42 children
  Interventions: Other: saliva

INTERVENTIONS:
Other: saliva — salivary secretion rate, salivary buffering capacity, pH, protein levels, superoxide dismutase (SOD), ferric reducing antioxidant power (FRAP), the thiobarbituric acid reactive substances (TBARS), protein carbonyl, protein thiols, total sialic acid.

SUMMARY:
The purpose of this study was to evaluate whether there are relationships between the salivary oxidative stress status of children with CHD directly dental caries including gender, age, salivary flow rate, salivary pH, salivary buffering capacity and drug intake such as angiotensin-converting enzyme (ACE) inhibitors. If such relationships exist, they might be employed to patient caries -prevention treatment.

DETAILED DESCRIPTION:
Using heart failure medications may cause low salivary pH and buffering capacity.As improved oral health is a priority for cardiac patients, it is necessary that they attend dental clinics for regular follow up.

This cross sectional study was carried out with 42 CHD and 42 healthy children who applied to Istanbul University, Faculty of Dentistry, Department of Pedodontics. Gender, age, general health and medications, and caries scores (dfs/DMFS) were recorded. Unstimulated saliva was collected from the participants and were assessed for the salivary secretion rate, salivary buffering capacity, pH, protein levels, superoxide dismutase (SOD), ferric reducing antioxidant power (FRAP), the thiobarbituric acid reactive substances (TBARS), protein carbonyl, protein thiols, total sialic acid.

ELIGIBILITY:
Inclusion Criteria:

* 3-12 years
* Caridac problems

Exclusion Criteria:

* other ages
* syndromes
* other systemic diseases

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2012-01-01 (Actual); Study Completion 2012-01-01 (Actual)

PRIMARY OUTCOMES:
salivary secretion rate | 2 hour
  salivary secretion rate
salivary buffering capacity | 2 hour
  salivary buffering capacity
pH | 2 hour
  pH

SECONDARY OUTCOMES:
protein levels of saliva | 2 hour
  protein levels
superoxide dismutase (SOD) | 2 hour
  superoxide dismutase (SOD)
ferric reducing antioxidant power (FRAP) | 2 hour
  ferric reducing antioxidant power (FRAP)
the thiobarbituric acid reactive substances (TBARS) | 2 hour
  the thiobarbituric acid reactive substances (TBARS)

OTHER OUTCOMES:
protein carbonyl | 2 hour
  protein carbonyl
protein thiols | 2 hour
  protein thiols
total sialic acid | 2 hour
  total sialic acid

IPD SHARING:
Plan to Share IPD: No